CLINICAL TRIAL: NCT07237867
Title: Frequency-Dependent Effects of Percutaneous Femoral Nerve Stimulation on Strength in Athletes With Patellar Tendinopathy: a Randomized Controlled Trial
Brief Title: Frequency-Dependent Effects of Percutaneous Femoral Nerve Stimulation on Quadriceps Strength in Athletes With Patellar Tendinopathy
Acronym: ppns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Xavier Picañol Parraga, Phd in Neuroscience, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-04-05
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Patellar Tendinopathy / Jumpers Knee
Keywords: Peripheral Percutaneous Nerve Stimulation; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Frequency PPNS (100 Hz) (Experimental): Participants receive peripheral percutaneous nerve stimulation (PPNS) applied to the femoral nerve at 100 Hz.
  Interventions: Device: Electrical stimulation
- Low-Frequency PPNS (2 Hz) (Experimental): Participants receive peripheral percutaneous nerve stimulation (PPNS) applied to the femoral nerve at 2 Hz.
  Interventions: Device: Electrical stimulation
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): Participants receive conventional transcutaneous electrical nerve stimulation (TENS) applied over the femoral nerve region using surface electrodes. Intensity is set at the maximal tolerated motor threshold to elicit visible quadriceps activation. The stimulation frequency and parameters are consistent with standard clinical practice for motor-level TENS.
  Interventions: Device: Electrical stimulation

INTERVENTIONS:
Device: Electrical stimulation — All electrical stimulation procedures are performed under real-time ultrasound guidance to accurately locate the femoral nerve and ensure safe and consistent electrode placement. For the percutaneous interventions (PPNS), a sterile needle electrode is inserted adjacent to the femoral nerve and stimulation is delivered at either high frequency (100 Hz) or low frequency (2 Hz), depending on the study arm. For the transcutaneous intervention (TENS), surface electrodes are positioned over the femoral nerve region using ultrasound guidance to confirm anatomical landmarks and optimize current delivery. In all conditions, stimulation is applied at the maximal tolerated motor threshold to elicit visible quadriceps activation.
  Other Names: Ultrasound-guided electrical stimulation

SUMMARY:
This study investigates the immediate effects of different peripheral electrical nerve stimulation protocols applied to the femoral nerve on quadriceps strength in athletes with patellar tendinopathy. Patellar tendinopathy is a common overuse injury that often reduces quadriceps activation and limits sports performance. Peripheral percutaneous nerve stimulation (PPNS) and transcutaneous electrical nerve stimulation (TENS) are frequently used in rehabilitation, but their frequency-dependent effects on muscle strength are not well established.

In this randomized crossover trial, each participant receives three stimulation protocols in separate sessions: high-frequency PPNS (100 Hz), low-frequency PPNS (2 Hz), and conventional TENS. All stimulation is delivered at the maximal tolerated motor threshold and, for PPNS conditions, under ultrasound guidance. Quadriceps maximal isometric strength is evaluated using an isometric force sensor before and after each intervention.

The primary objective is to compare the acute changes in maximal voluntary contraction (MVC) following each stimulation protocol. The study aims to clarify whether different stimulation frequencies can enhance, reduce, or have no effect on quadriceps strength in this athletic population.

By identifying frequency-specific neuromodulatory responses, this study may help clinicians and sports practitioners select the most appropriate stimulation parameters to optimize rehabilitation and performance in individuals with patellar tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 40 years.
* Recreational or competitive athletes with clinically diagnosed patellar tendinopathy for at least 3 months.
* Ultrasound-confirmed patellar tendinopathy, including hypoechoic areas, tendon thickening, or neovascularization consistent with clinical diagnosis.

Presence of pain during tendon-loading activities (e.g., jumping, running, squatting).

* Ability to perform maximal voluntary isometric contractions of the quadriceps.
* Ability to comply with all study procedures and attend all experimental sessions.
* Written informed consent obtained prior to participation.

Exclusion Criteria:

* Previous knee surgery or traumatic knee injury within the past 12 months.
* Complete or partial patellar tendon rupture.
* Neurological disorders affecting lower limb strength or motor control.
* Contraindications to electrical stimulation, including implanted electrical devices (e.g., pacemaker).
* Current lower-limb radiculopathy or neuropathy.
* Skin infections, open wounds, or dermatological conditions at the stimulation site.
* Use of analgesics, anti-inflammatories, or corticosteroid injections within the past 48 hours.
* Participation in another interventional study in the previous 30 days.
* Pregnancy or suspected pregnancy.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Quadriceps Maximal Isometric Voluntary Contraction (MVC) | Baseline (pre-intervention), and at 2 minutes, 10 minutes, 15 minutes, and 30 minutes post-intervention.
  Quadriceps maximal isometric voluntary contraction (MVC) is measured using a calibrated isometric force sensor with the participant seated and the knee positioned at 60° of flexion. MVC is recorded as the peak force output during a standardized 5-second maximal contraction. The primary endpoint is the change in MVC from pre-intervention to immediately post-intervention across the three stimulation conditions (high-frequency PPNS, low-frequency PPNS, and TENS). Higher values indicate greater quadriceps force production.

SECONDARY OUTCOMES:
Change in Quadriceps Rate of Force Development (RFD 0-250 ms) | Baseline (pre-intervention), and at 2 minutes, 10 minutes, 15 minutes, and 30 minutes post-intervention.
  Quadriceps rate of force development (RFD) in the early phase of contraction (0-250 ms) is calculated from the force-time curve obtained during maximal isometric voluntary contractions using a calibrated isometric force sensor. RFD 0-250 ms reflects the participant's ability to rapidly generate force and is derived as the slope of the force increase within the first 250 milliseconds. The outcome measure is the change in RFD between baseline and the post-intervention time points across the three stimulation conditions (high-frequency PPNS, low-frequency PPNS, and TENS).
Change in Quadriceps Impulse (0-250 ms) | Baseline (pre-intervention), and at 2 minutes, 10 minutes, 15 minutes, and 30 minutes post-intervention.
  Quadriceps impulse (0-250 ms) is calculated as the integrated area under the force-time curve during the first 250 milliseconds of a maximal isometric voluntary contraction, recorded using a calibrated isometric force sensor. This metric reflects the combined ability to rapidly generate and sustain force during the early phase of contraction. The outcome measure is the change in impulse between baseline and post-intervention assessments across the three stimulation conditions (high-frequency PPNS, low-frequency PPNS, and TENS).
Incidence of Adverse Events Assessed Through Post-Intervention Questionnaires | Immediately after each intervention session.
  Adverse events related to the stimulation procedures are assessed using a standardized post-intervention questionnaire completed immediately after each stimulation session. Participants are asked to report the presence and severity of any undesirable effects, including discomfort, pain, bleeding, bruising, transient paresthesia, dizziness, or any unexpected symptoms. All adverse events are recorded, categorized by type and severity, and evaluated for their potential relationship to the intervention (high-frequency PPNS, low-frequency PPNS, or TENS). No serious adverse events are anticipated due to the low-risk nature of the procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Blanquerna University, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
No final decision has yet been made regarding the sharing of de-identified individual participant data (IPD) from this study. Data sharing may be considered after publication of the study results and pending compliance with ethical approvals, institutional policies, and participant confidentiality protections. Only fully de-identified datasets would be eligible for potential sharing.
  Access Criteria and How to Request IPD
  If data sharing is approved in the future, de-identified IPD will be made available to qualified researchers upon reasonable request. Interested investigators may contact the Principal Investigator with a methodologically sound proposal. Access will be granted only after review of the request and signature of a data use agreement.